CLINICAL TRIAL: NCT02565134
Title: Multi Center, Double-blind, Randomized, Placebo-controlled Parallel-group, Dose Finding Phase II Clinical Trial to Evaluate Antipruritic Effect and Safety of PAC-14028 Cream (0.1%, 0.3%, 1.0%) in Skin Pruritus Patients
Brief Title: A Study to Evaluate the Safety and Efficacy of PAC-14028 Cream in Skin Pruritus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP-TRPV1_PII-02
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Skin Pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PAC-14028 cream 0.1% (Experimental): PAC-14028 cream 0.1%, Twice daily for 4 weeks
  Interventions: Drug: PAC-14028 cream 0.1%
- PAC-14028 cream 0.3% (Experimental): PAC-14028 cream 0.3%, Twice daily for 4 weeks
  Interventions: Drug: PAC-14028 cream 0.3%
- PAC-14028 cream 1.0% (Experimental): PAC-14028 cream 1.0%, Twice daily for 4 weeks
  Interventions: Drug: PAC-14028 cream 1.0%
- PAC-14028 cream vehicle (Placebo Comparator): PAC-14028 cream vehicle, Twice daily for 4 weeks
  Interventions: Drug: PAC-14028 cream vehicle

INTERVENTIONS:
Drug: PAC-14028 cream 0.1% — Topical application
  Arms: PAC-14028 cream 0.1%
Drug: PAC-14028 cream 0.3% — Topical application
  Arms: PAC-14028 cream 0.3%
Drug: PAC-14028 cream 1.0% — Topical application
  Arms: PAC-14028 cream 1.0%
Drug: PAC-14028 cream vehicle — Topical application
  Arms: PAC-14028 cream vehicle

SUMMARY:
The study is a Phase II, multi center, randomized, double-blind, placebo-controlled study in male and female subjects, aged ≥ 19 years with skin pruritus. All subjects will receive BID topical applications of PAC-14028 cream or vehicle for up to 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 19 - 70 years
* Patients who have eczema or xerosis cutis at the area where investigational product is applied (arm or leg)
* Patients whose result of the pruritus test (Visual Analogue Scale, VAS) at Visit 1 and 2 is 5 or more
* Patients whose overall dry skin score of the area where investigational product is applied at Visit 1 and 2 is 2 points or more

Exclusion Criteria:

* Patients with pruritus caused by other medical, psychotic and nervous causes other than the skin disease
* Patients with such skin diseases as malignant tumor or chronic urticaria among patients with skin diseases
* Patients with simple pruritus caused by such allergic material as scabies, and insect bite wound
* Patients with the symptom of systemic infection at the time of the participation in the clinical study
* Patients with a history of taking topical treatment drug, topical steroid agent or antibiotics for the treatment of pruritus within 2 weeks
* Patients with a history of taking oral steroid agent within 4 weeks
* Patients with a history of taking a physical treatment for the treatment of pruritus including phototherapy within 4 weeks
* Pregnant or breast-feeding women
* Women at a childbearing age who has childbearing potential or has a plan to get pregnant during the clinical study period

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in intensity of pruritus as measured by 10 cm VAS | Week 4 from baseline

SECONDARY OUTCOMES:
Treatment success rate (A decrease in VAS by 2 or more is judged as a success) | Week 4 from baseline
Change in Overall Dry Skin (ODS) score | Week 4 from baseline
Change in Transepidermal Water Loss (TEWL) | Week 4 from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Miyoung Park, PhD, Study Director — Amorepacific R&D Center
Locations (1):
- Seoul National University Hospital, Seoul, South Korea